CLINICAL TRIAL: NCT06032910
Title: The Use of Surgical Mesh in Open Radical Cystectomy With Ileal Conduit Urinary Diversion to Prevent Parastomal Hernias
Brief Title: Surgical Mesh in Radical Cystectomy to Prevent Parastomal Hernias
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mesh_RACE
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Bladder Cancer; Hernia; Ileal Conduit
Keywords: radical cystectomy; ileal conduit; parastomal hernia; mesh
MeSH Terms: conditions — Urinary Bladder Neoplasms; Hernia | interventions — Surgical Mesh

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Patients who receive prophylactic mesh during the surgery.
  Interventions: Device: Surgical mesh

INTERVENTIONS:
Device: Surgical mesh — Prophylactic synthetic non-absorbable keyhole mesh placement upon construction of ileal conduit.

SUMMARY:
Radical cystectomy with ileal conduit urinary diversion serves as a foundational curative treatment strategy for selected patients afflicted with urothelial carcinoma of the bladder. Parastomal hernia after this procedure is an underestimated and undertreated clinical entity, which heavily impairs patients' quality of life due to symptoms of pain, leakage, application or skin problems. There is little evidence about prophylactic mesh placement for parastomal hernia prevention. In this study we examine the use of meshes during radical cystectomy and compare them with a control group.

DETAILED DESCRIPTION:
Radical cystectomy with ileal conduit diversion is a procedure possible with complications. A primary stoma-related complication is the parastomal hernia (PH), which presents significant challenges to both the medical community and the patient. PH is classically defined as the protrusion of abdominal contents via the abdominal wall, especially in the direct vicinity of a stoma, whether it be a colostomy, ileostomy, or ileal conduit stoma. The incidence of PH post ileal conduit urinary diversion is especially concerning, with reports estimating its occurrence at around 17%. This data only emphasizes the need to reevaluate and optimize surgical treatments for PH, particularly as, in many cases, management strategies are extrapolated from experiences with colostomies or ileostomies. Notably, PHs are often described after these procedures rather than RC with ileal conduit urinary diversion. Further complicating the issue is the fact that estimates suggest around 30% of patients develop a PH within 12 months post any type of stoma site surgery. For those undergoing ileal conduit urinary diversion specifically, recurrence rates following PH repair can be alarmingly high, with figures as steep as 69% within a year.

ELIGIBILITY:
Inclusion Criteria:

* muscle-invasive or high-risk non-muscle-invasive bladder cancer patients

Exclusion Criteria:

* different than surgical therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Parastomal hernia | 12 months
  Incidence after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Department's website — https://www.fnhk.cz/urol